CLINICAL TRIAL: NCT04430751
Title: Medical Qigong for Mobility and Balance Self-Confidence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, James E. Stahl, MD, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 250-37
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Falls, Balance Self-confidence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate start (Active Comparator)
  Interventions: Behavioral: Medical QiGong training
- wait time control (Active Comparator)
  Interventions: Behavioral: Medical QiGong training

INTERVENTIONS:
Behavioral: Medical QiGong training — The study intervention consisted of a 12-week training program that introduced students to a progressive series of 10 QiGong "forms" that are designed to build upon each other to restore balance and function and to enhance well-being. These forms involve both physical movement and visualization.

SUMMARY:
The population is aging and increasingly at risk for falls and fractures with substantial consequences to wellbeing, health and costs. Training interventions such as Tai Chi have been demonstrated to help reduce these risks. Tai chi is a subset of both martial and medical qi gong.

This is a prospective intervention study with wait time control that will examine the ability of a manualized medical qi gong training protocol improve balance, gait and health self-confidence.

The intervention is a 12 week manualized medical qi gong training program where students are taught a progressive series of 10 qi gong forms that are designed to build upon each other and restore balance and function. These forms involve both physical movement and visualization.

The Community Balance and Mobility scale (a performance based measure) and Activities-specified Balance Confidence scale (a survey)will be the prime outcome instruments

ELIGIBILITY:
Inclusion Criteria:

* Adults 50 years of age or older who presented at the two study locations (Massachusetts, Arizona) were considered eligible for participation

Exclusion Criteria:

* Unable to participate in informed consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Community Balance and Mobility Scale | through study completion, up to 16 weeks

SECONDARY OUTCOMES:
Activities-specific Balance Confidence Scale | through study completion, up to 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Yes
blinded de-identified information will be shared at request
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Stahl JE, Belisle SS, Zhao W. Medical Qigong for Mobility and Balance Self-Confidence in Older Adults. Front Med (Lausanne). 2020 Aug 14;7:422. doi: 10.3389/fmed.2020.00422. eCollection 2020. PMID 32923446